CLINICAL TRIAL: NCT03767621
Title: Concordance Between FFR and iFR for the Assessment of Intermediate Lesions in the Left Main Coronary Artery. A Prospective Validation of a Default Value for iFR (iLITRO Study)
Brief Title: Concordance Between FFR and iFR for the Assessment of Intermediate Lesions in the Left Main Coronary Artery. A Prospective Validation of a Default Value for iFR
Acronym: iLITRO
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: iLITRO EPIC-07
Record Dates: First submitted 2018-12-02; First posted 2018-12-06 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease; Left Main Coronary Artery Stenosis; Left Main Coronary Artery Disease; Restenosis, Coronary
Keywords: Left Main Coronary Artery; Intermediate Coronary Lesions; iFR; Coronary Physiology; IVUS
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with intermediate lesions.: Patients with intermediate lesions (stenosis in angiography between 25% and 60%) in LMCA.
  Interventions: Other: Indication of revascularization

INTERVENTIONS:
Other: Indication of revascularization — Device: iFR/FFR

SUMMARY:
The assessment of Left Main Coronary Artery (LMCA) lesions by means of coronary angiography renders serious limitations.

Studies with a limited number of patients have shown that a value of FFR (Fractional Flow Reserve) above 0.80 identify a low risk of events in case of not performing revascularization in patients with intermediate stenosis in the LMCA. Although iFR (Instant wave Free Ratio) has recently been found equivalent to FFR The demonstration of the prognostic utility of iFR in patients with LMCA intermediate lesions could have an important clinical impact and justify its systematic use for the treatment decision in these high-risk patients.

DETAILED DESCRIPTION:
The assessment of Left Main Coronary Artery (LMCA) lesions by means of coronary angiography renders serious limitations. In the case of intermediate stenoses (25-60%), invasive imaging tests, intravascular ultrasound (IVUS) or optical coherence tomography (OCT) or functional by determining the Fractional Flow Reserve (FFR), have been proposed to identify those patients who could benefit from revascularization.

Studies with a limited number of patients have shown that a value of FFR above 0.80 identify a low risk of events in case of not performing revascularization in patients with intermediate stenosis in the LMCA. Although iFR (Instant wave Free Ratio) has recently been found equivalent to FFR in assessing the prognosis of patients with intermediate lesions, the validation of the prognostic power of this index in patients with intermediate LMCA lesions has not been demonstrated, although it is used in clinical practice assuming the results in other locations of the lesions.

The demonstration of the prognostic utility of iFR in patients with LMCA intermediate lesions could have an important clinical impact and justify its systematic use for the treatment decision in these high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermediate lesion in the LMCA (25-60% angiographic stenosis) by visual estimation) in which the realization of a study with guide of pressure for the determination of the iFR.
* Patients aged ≥18 years.
* Patients able of giving informed consent.

Exclusion Criteria:

* Patients with indication for coronary surgery regardless of the significance of the LMCA lesion.
* Patients with a LMCA lesion presenting with ulceration, dissection or thrombus.
* Patients with previous arterial or venous graft lesion functioning in the territory irrigated by the LMCA (LMCA protected).
* Patients with ACS (Acute Coronary Syndrome) with a potentially guilty lesion in the LMCA.
* Patients unable to obtain informed consent.
* Patients with known terminal illness that conditions a life expectancy less than 1 year.
* Patients with hemodynamic instability with Killip III or IV class.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate stenosis of the LMCA will be included by coronary angiography (estimate visual 25-60%) in which a functional study is performed with pressure and calculation guidance of iFR and FFR with intravenous adenosine in perfusion to guide the indication of revascularization.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessment correlation between FFR>=0.80 and iFR >=0.89 | 1 day
  Efficacy and correlation of two invasive indexes of functional assessment by intracoronary pressure guidance in intermediate lesions of the LMCA with a cut-off point to defer the treatment of FFR> = 0.80 (with intravenous adenosine) and iFR > = 0.89. the LMCA.
Major Adverse Cardiac Events | 30 days
  Composite of death, myocardial infarction, unplanned revascularisation
Major Adverse Cardiac Events | 1 year
  Composite of death, myocardial infarction, unplanned revascularisation
Major Adverse Cardiac Events | 5 years
  Composite of death, myocardial infarction, unplanned revascularisation

SECONDARY OUTCOMES:
Assessment correlation between iFR and IVUS | 5 years
  Assessment correlation between iFR and IVUS derived minimal luminal area
Death (all cause) | 30 days, 1 and 5 years
  Death (all cause)
Death (cardiovascular) | 30 days, 1 and 5 years
  Death (cardiovascular)
Non-fatal Myocardial Infarction | 30 days, 1 and 5 years
  Non-fatal Myocardial Infarction
Non-fatal Myocardial Infarction related to the LMCA lesion | 30 days, 1 and 5 years
  Non-fatal Myocardial Infarction related to the LMCA lesion
Revascularization | 30 days, 1 and 5 years
  Revascularization
Revascularization of the target lesion | 30 days, 1 and 5 years
  Revascularization of the target lesion
Myocardial Infarction related to target lesion revascularization | 30 days, 1 and 5 years
  Myocardial Infarction related to target lesion revascularization
Stent Thrombosis in the target lesion revascularization | 30 days, 1 and 5 years
  Stent Thrombosis in the target lesion revascularization
Restenosis of the stent in target lesion | 30 days, 1 and 5 years
  Restenosis of the stent in target lesion
New revascularization of the target lesion | 30 days, 1 and 5 years
  New revascularization of the target lesion

CONTACTS AND LOCATIONS:
Overall Officials: José María de la Torre, PhD, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla; Oriol Rodríguez Leor, PhD, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (38):
- Spain (38):
  - Hospital Universitari Mutua de Terrassa, Terrassa, Barcelona
  - Hospital General Universitario de Santa Lucia de Cartagena, Cartagena, Murcia
  - Hospital Clinico Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Hospital General Universitario de Castellón, Castellon, Valencia
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya
  - Hospital General Universitario de Albacete, Albacete
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitari Germans Trias I Pujol de Badalona, Badalona
  - Hospital Del Mar, Barcelona
  - Hospital Clinic I Provincial de Barcelona, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Bellvitge, Barcelona
  - Hospital Universitario Puerto Real, Cadiz
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitari Doctor Josep Trueta, Girona
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital General Juan Ramón Jiménez, Huelva
  - Hospital de León, León
  - Hospital Universitari Lucus Agusti, Lugo
  - Hospital de La Princesa, Madrid
  - Clinica Universitaria de Navarra, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital de Merida, Mérida
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitari Joan Xxiii de Tarragona, Tarragona
  - Hospital Universitario Virgen de La Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari I Politecnic La Fe, Valencia
  - Hospital Universitario Alvaro Cunqueiro, Vigo
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] De Bruyne B, Baudhuin T, Melin JA, Pijls NH, Sys SU, Bol A, Paulus WJ, Heyndrickx GR, Wijns W. Coronary flow reserve calculated from pressure measurements in humans. Validation with positron emission tomography. Circulation. 1994 Mar;89(3):1013-22. doi: 10.1161/01.cir.89.3.1013. PMID 8124786
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Pijls NH, van Schaardenburgh P, Manoharan G, Boersma E, Bech JW, van't Veer M, Bar F, Hoorntje J, Koolen J, Wijns W, de Bruyne B. Percutaneous coronary intervention of functionally nonsignificant stenosis: 5-year follow-up of the DEFER Study. J Am Coll Cardiol. 2007 May 29;49(21):2105-11. doi: 10.1016/j.jacc.2007.01.087. Epub 2007 May 17. PMID 17531660
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] Sen S, Escaned J, Malik IS, Mikhail GW, Foale RA, Mila R, Tarkin J, Petraco R, Broyd C, Jabbour R, Sethi A, Baker CS, Bellamy M, Al-Bustami M, Hackett D, Khan M, Lefroy D, Parker KH, Hughes AD, Francis DP, Di Mario C, Mayet J, Davies JE. Development and validation of a new adenosine-independent index of stenosis severity from coronary wave-intensity analysis: results of the ADVISE (ADenosine Vasodilator Independent Stenosis Evaluation) study. J Am Coll Cardiol. 2012 Apr 10;59(15):1392-402. doi: 10.1016/j.jacc.2011.11.003. Epub 2011 Dec 7. PMID 22154731
- [Background] Davies JE, Sen S, Dehbi HM, Al-Lamee R, Petraco R, Nijjer SS, Bhindi R, Lehman SJ, Walters D, Sapontis J, Janssens L, Vrints CJ, Khashaba A, Laine M, Van Belle E, Krackhardt F, Bojara W, Going O, Harle T, Indolfi C, Niccoli G, Ribichini F, Tanaka N, Yokoi H, Takashima H, Kikuta Y, Erglis A, Vinhas H, Canas Silva P, Baptista SB, Alghamdi A, Hellig F, Koo BK, Nam CW, Shin ES, Doh JH, Brugaletta S, Alegria-Barrero E, Meuwissen M, Piek JJ, van Royen N, Sezer M, Di Mario C, Gerber RT, Malik IS, Sharp ASP, Talwar S, Tang K, Samady H, Altman J, Seto AH, Singh J, Jeremias A, Matsuo H, Kharbanda RK, Patel MR, Serruys P, Escaned J. Use of the Instantaneous Wave-free Ratio or Fractional Flow Reserve in PCI. N Engl J Med. 2017 May 11;376(19):1824-1834. doi: 10.1056/NEJMoa1700445. Epub 2017 Mar 18. PMID 28317458
- [Background] Gotberg M, Christiansen EH, Gudmundsdottir IJ, Sandhall L, Danielewicz M, Jakobsen L, Olsson SE, Ohagen P, Olsson H, Omerovic E, Calais F, Lindroos P, Maeng M, Todt T, Venetsanos D, James SK, Karegren A, Nilsson M, Carlsson J, Hauer D, Jensen J, Karlsson AC, Panayi G, Erlinge D, Frobert O; iFR-SWEDEHEART Investigators. Instantaneous Wave-free Ratio versus Fractional Flow Reserve to Guide PCI. N Engl J Med. 2017 May 11;376(19):1813-1823. doi: 10.1056/NEJMoa1616540. Epub 2017 Mar 18. PMID 28317438
- [Background] de la Torre Hernandez JM, Hernandez Hernandez F, Alfonso F, Rumoroso JR, Lopez-Palop R, Sadaba M, Carrillo P, Rondan J, Lozano I, Ruiz Nodar JM, Baz JA, Fernandez Nofrerias E, Pajin F, Garcia Camarero T, Gutierrez H; LITRO Study Group (Spanish Working Group on Interventional Cardiology). Prospective application of pre-defined intravascular ultrasound criteria for assessment of intermediate left main coronary artery lesions results from the multicenter LITRO study. J Am Coll Cardiol. 2011 Jul 19;58(4):351-8. doi: 10.1016/j.jacc.2011.02.064. PMID 21757111
- [Background] Hamilos M, Muller O, Cuisset T, Ntalianis A, Chlouverakis G, Sarno G, Nelis O, Bartunek J, Vanderheyden M, Wyffels E, Barbato E, Heyndrickx GR, Wijns W, De Bruyne B. Long-term clinical outcome after fractional flow reserve-guided treatment in patients with angiographically equivocal left main coronary artery stenosis. Circulation. 2009 Oct 13;120(15):1505-12. doi: 10.1161/CIRCULATIONAHA.109.850073. Epub 2009 Sep 28. PMID 19786633
- [Background] de la Torre Hernandez JM, Baz Alonso JA, Gomez Hospital JA, Alfonso Manterola F, Garcia Camarero T, Gimeno de Carlos F, Roura Ferrer G, Recalde AS, Martinez-Luengas IL, Gomez Lara J, Hernandez Hernandez F, Perez-Vizcayno MJ, Cequier Fillat A, Perez de Prado A, Gonzalez-Trevilla AA, Jimenez Navarro MF, Mauri Ferre J, Fernandez Diaz JA, Pinar Bermudez E, Zueco Gil J; IVUS-TRONCO-ICP Spanish study. Clinical impact of intravascular ultrasound guidance in drug-eluting stent implantation for unprotected left main coronary disease: pooled analysis at the patient-level of 4 registries. JACC Cardiovasc Interv. 2014 Mar;7(3):244-54. doi: 10.1016/j.jcin.2013.09.014. PMID 24650399
- [Derived] Rodriguez-Leor O, de la Torre Hernandez JM, Garcia-Camarero T, Garcia Del Blanco B, Lopez-Palop R, Fernandez-Nofrerias E, Cuellas Ramon C, Jimenez-Kockar M, Jimenez-Mazuecos J, Fernandez Salinas F, Gomez-Lara J, Brugaletta S, Alfonso F, Palma R, Gomez-Menchero AE, Millan R, Tejada Ponce D, Linares Vicente JA, Ojeda S, Pinar E, Fernandez-Pelegrina E, Morales-Ponce FJ, Cid-Alvarez AB, Rama-Merchan JC, Molina Navarro E, Escaned J, Perez de Prado A. Instantaneous Wave-Free Ratio for the Assessment of Intermediate Left Main Coronary Artery Stenosis: Correlations With Fractional Flow Reserve/Intravascular Ultrasound and Prognostic Implications: The iLITRO-EPIC07 Study. Circ Cardiovasc Interv. 2022 Nov;15(11):861-871. doi: 10.1161/CIRCINTERVENTIONS.122.012328. Epub 2022 Sep 16. PMID 36111801